CLINICAL TRIAL: NCT04834336
Title: Effects of Inspiratory Muscle Training in Patients With Acute Decompensated Heart Failure
Brief Title: Inspiratory Muscle Training in Acute Decompensated Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Aylin Tanriverdi, Research assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5883-GOA
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical training plus inspiratory muscle training (Experimental): Inspiratory Muscle Training (IMT) will be implemented by using the Power Breathe® device. IMT training will begin with mild to moderate intensity of maximal inspiratory pressure. It will be performed 6 to 10 breaths, 4 sets, and twice daily during the hospitalization when as soon as hemodynamic stability is provided.
  Physical Training will consist of each functional domain (balance, mobility, strength, and endurance) according to patients' functional levels. These will include static and dynamic balance training, mobility training, functional strength training focused on lower extremities, and endurance training as sustained walking. A daily 30 min session during the hospitalization will be performed with one-on-one supervision when as soon as hemodynamic stability is provided.
  Interventions: Device: inspiratory muscle training device; Other: Physical training
- Physical training (Active Comparator): Physical Training will consist of each functional domain (balance, mobility, strength, and endurance) according to patients' functional levels. These will include static and dynamic balance training, mobility training, functional strength training focused on lower extremities, and endurance training as sustained walking. A daily 30 min session during the hospitalization will be performed with one-on-one supervision when as soon as hemodynamic stability is provided.
  Interventions: Other: Physical training

INTERVENTIONS:
Device: inspiratory muscle training device — Inspiratory muscle training will be performed with an inspiratory muscle training device.
  Arms: Physical training plus inspiratory muscle training
Other: Physical training — Physical training will be performed with exercise including balance, mobility, functional strength, and endurance.

SUMMARY:
Hospitalized patients with acute decompensated heart failure (ADHF) present a high prevalence of inspiratory muscle weakness on admission and discharge. Inspiratory muscle training has been reported as a beneficial approach in chronic heart failure. However, the effects of inspiratory muscle training in hospitalized patients with ADHF have been not known. The aim of this study is to investigate the safety, feasibility, and effects of inspiratory muscle training in hospitalized patients with ADHF.

DETAILED DESCRIPTION:
The participants will randomly be allocated into two groups: (1) Physical training plus inspiratory muscle training, (2) Physical training

Participants in the physical training plus inspiratory muscle training group will perform inspiratory muscle training and physical training. Inspiratory muscle training will be applied with an electronic device. Physical training will be implemented as balance, mobility, functional strength, endurance exercises. During the hospitalization, the inspiratory muscle training will be carried out twice a day with mild to moderate whereas physical training will be carried out once a day. The physical training group will perform only physical training. Physical training will be implemented as balance, mobility, functional strength, endurance exercises. During the hospitalization, physical training will be carried out once a day. For the safety and feasibility of inspiratory muscle training, data will be collected daily during the hospitalization. For effects of inspiratory muscle training, data will be collected at baseline and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* The management of a diagnosis of ADHF over 24 hours in a hospital setting
* Hemodynamic stability
* The independence of basic activities of daily life before admission

Exclusion Criteria:

* Acute myocardial infarction
* Congenital heart disease
* Endocarditis, miyocarditis or pericarditis
* Morbid obesity
* Already participating in cardiac rehabilitation

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | baseline and hospital discharge, an average of 4 to 10 days
  Maximal inspiratory pressure will be measured by an electronic mouth pressure device (cmH2O)

SECONDARY OUTCOMES:
Adverse events | During the hospitalization, daily, during an average of 4 to 10 days
  The number of adverse events resulting from the intervention will be noted. Adverse events include blood pressure greater than 170/100 mmHg, desaturation of oxygen greater than 4%, severe musculoskeletal and/or chest pain, dyspnea greater than 6 on the Borg scale, dizziness, nausea, vomiting, bleeding, loss or obstruction of the central or peripheral catheter.
Recruitment rate | During the hospitalization, daily, during an average of 4 to 10 days
  The number of participants divided by the total number of eligible patients (%)
Adherence rate | During the hospitalization, daily, during an average of 4 to 10 days
  The number of training sessions divided by the total number of potential sessions (%)
Retention rate | During the hospitalization, daily, during an average of 4 to 10 days
  The number of patients who complete the protocol divided by the total number of patients included in the study (%)
New York Heart Association Functional Classification | baseline and hospital discharge, an average of 4 to 10 days
  Functional Classification will be assessed with New York Heart Association (NYHA) Functional Classification. The minimum value is 1 whereas the maximum value is 4. Higher scores indicate the lower functional class.
Dyspnea | baseline and hospital discharge, an average of 4 to 10 days
  Dyspnea will be assessed by using the Modified Medical Research Council Scale. It is a 5-item scale. Higher scores indicate higher dyspnea perception.
Hand Grip Strength | baseline and hospital discharge, an average of 4 to 10 days
  Hand grip strength will be measured by a dynamometer.
Physical Performance | baseline and hospital discharge, an average of 4 to 10 days
  Physical performance will be measured by Short Physical Performance Battery (SPPB). SPPB comprises 5 times sit-to-stand, standing balance and 4-m gait speed. The total score ranges from 0 to 12 and a higher score indicates better physical performance.
Frailty | baseline and hospital discharge, an average of 4 to 10 days
  Frailty will be assessed by using the Clinical Frailty Scale (CFS). CFS scores on a scale from 1 (very fit) to 9 (terminally ill).
Cardiac autonomic function | baseline and hospital discharge, an average of 4 to 10 days
  Cardiac autonomic function will be evaluated with heart rate variability analysis by using a SphygmoCor ® device.
Arterial Stiffness | baseline and hospital discharge, an average of 4 to 10 days
  Arterial stiffness will be measured by augmentation index using a SphygmoCor® device.
Disability | baseline and hospital discharge, an average of 4 to 10 days
  Disability will be assessed by using Barthel Index. It occurs 10 questions and the score ranges from 0 to 100. Higher scores indicate greater independence.
One-year mortality | one year after discharge
  The mortality rate during the first year following hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sema Savci, Prof, Study Director — Dokuz Eylul University

IPD SHARING:
Plan to Share IPD: No